CLINICAL TRIAL: NCT05027958
Title: Characterization of Tissue-Specific Immune Responses to Bronchoscopic Instillation of Mycobacterial Antigens Into the Human Lung
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 210027; 21-H-0027
Record Dates: First submitted 2021-08-28; First posted 2021-08-31 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-01-16

CONDITIONS: Healthy; Latent Tuberculosis Infection (LTBI)
Keywords: Tuberculin Purified Protein Derivative; PPD; antigen-specific immune cells in airways
MeSH Terms: conditions — Latent Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Healthy Volunteer Participants with confirmed Latent Tuberculosis Infection (LTBI) (Other): Healthy volunteer participants with confirmed Latent Tuberculosis Infection (LTBI) (TST positive and IGRA positive) receiving instillation dose of purified protein derivative (PPD) 0.5 tuberculin units (10 uL Tubersol® in 10 mL normal saline) into the right upper lobe of lung.
  Interventions: Drug: Tuberculin Purified Protein Derivative
- Arm 2: Healthy Volunteer Participants with confirmed non-Latent Tuberculosis Infection (LTBI) (Other): Healthy volunteer participants with confirmed non-Latent Tuberculosis Infection (LTBI) (TST negative and IGRA negative) receiving instillation dose of purified protein derivative (PPD) 0.5 tuberculin units (10 uL Tubersol® in 10 mL normal saline) into the right upper lobe of lung.
  Interventions: Drug: Tuberculin Purified Protein Derivative

INTERVENTIONS:
Drug: Tuberculin Purified Protein Derivative — PPD administered through the airways to elicit the development of alveolar inflammation challenge dose of 0.5 TU

SUMMARY:
Background:

Tuberculosis (TB) is a lung disease. It is caused by inhaling a type of airborne bacterium. Tuberculin Purified Protein Derivative (PPD) is used to test for TB exposure. It is usually injected under a person s skin. In this study, it will be applied in the lung.

Objective:

To learn how the cells within the lung react (immune response) when exposed to PPD.

Eligibility:

Adults ages 18-64 who (1) have been exposed to TB but do not have active disease or symptoms or (2) have never been exposed to TB.

Design:

Participants will be screened with a medical history, physical exam, and blood tests. They will have a TB skin test. They will also have an electrocardiogram to examine heart rhythm. For this, sticky patches will be placed on their chest.

Some screening tests will be repeated at study visits.

Participants will have 3 FDG PET-CT scans. They will lie in a machine that creates pictures of the inside of their body. They will get a radioactive substance injected into their arm called 18FDG. It helps make the pictures.

Participants will have 3 bronchoscopies. Their mouth and nasal airways will be numbed. They will get drugs to relax. A tube will be inserted through their nose or mouth into a lung. Fluid will be delivered into the lung and suctioned back out to collect cells. They will get PPD during the first bronchoscopy.

Participation will last for about 30 days. Participants will visit the clinic up to 8 times. They will go home after each procedure. No hospital stays are needed....

DETAILED DESCRIPTION:
Study Description: We propose a pilot study in which we employ directed bronchoscopic instillation of Mycobacterium tuberculosis (Mtb)-Tuberculin Purified Protein Derivative (PPD) to evaluate local airway immune response in adults with or without latent tuberculosis infection (LTBI).

Primary Objective: The primary objective of this study is to understand the pulmonary immune response to mycobacterial antigens by determining the persistence of antigen-specific immune cells in the airways versus circulation after local bronchoscopic instillation of Tuberculin Purified Protein Derivative (PPD) into the lungs of adults with or without LTBI.

Secondary Objective: The secondary objective is to characterize the location and persistence of immune cell activity in the pulmonary parenchyma and thoracic lymph nodes with positron emission tomography combined with chest computed tomography (PET-CT) after bronchoscopic Tuberculin Purified Protein Derivative (PPD) instillation in adults with or without LTBI.

Exploratory Objectives: (a) An exploratory objective will be to perform phenotypic and functional analysis of immune cell populations in the airways vs circulation following bronchoscopic instillation of Tuberculin Purified Protein Derivative (PPD) into the lungs of individuals with or without LTBI. (b) An additional exploratory objective will be to characterize the production of soluble mediators (including but not limited to: cytokines, lipid mediators, and defensins) in BAL fluid vs blood within the same context.

Endpoints:

Primary Endpoint: The primary endpoint will be the enumeration of Mtb antigen-specific CD4+ and CD8+ T cell populations in the airway and peripheral blood at early and late time points after bronchoscopic Tuberculin Purified Protein Derivative (PPD) instillation.

Secondary Endpoint: The secondary endpoint will be the quantification of [18F]fluoro-D-glucose (FDG) uptake in adjacent pulmonary parenchyma and draining thoracic lymph nodes via PET-CT at early and late time points after PPD instillation.

Exploratory Endpoints: (a) An exploratory endpoint will be the quantification of frequencies of cell surface molecules, intracellular cytokines and transcription factors among immune cell populations in the airways vs circulation following bronchoscopic instillation of Tuberculin Purified Protein Derivative (PPD) into the lungs of individuals with or without LTBI. (b) An exploratory endpoint will involve the identification and quantification of soluble mediators in the airway and peripheral blood after PPD instillation in the lungs within the same context.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults 18-64 years old will be recruited for the two groups (non-LTBI controls vs confirmed LTBI). The lower limit of this age range is based on the need for invasive bronchoscopic procedures and exposure to radiation, both of which carry more risk at younger ages. In addition, most adults present with post-primary or reactivation TB that most often occurs radiographically in the upper lobes of the lungs, often with cavitation. Conversely, children and rare adults with primary TB have non-cavitary disease in the lower lobes. The higher limit of this age range is based on the known property of immune senescence, i.e., the waning of the strength of immune responses with advancing age.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 - 64 years of age
* No significant active medical problems. This would include but not limited to any cardiac disorder (e.g. arrhythmia, valvular disease), pulmonary disease (e.g. asthma requiring chronic medications, chronic bronchitis, emphysema, obstructive sleep apnea), kidney disease (e.g. nephritis, nephrosis), rheumatologic disorder (e.g. inflammatory arthritis), endocrine disorder (e.g. diabetes, thyroid disease), liver disease (e.g. hepatitis), gastrointestinal disorder (e.g. inflammatory bowel disease) or infectious disease (e.g. active tuberculosis).
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and agreement to use such a method during study participation

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy as assessed by urinary or plasma HCG or breastfeeding
* History of clinically significant respiratory dysfunction 3 months prior to participating

  * Evidence of new pulmonary infection
  * History of any chronic lung infections or chronic lung disease
  * History of pulmonary hypertension
  * Need for supplemental oxygen administration at rest
* Current use or inability to suspend use of anticoagulant therapy including platelet inhibitors (e.g. clopidogrel) within 7 days of study bronchoscopy or systemic anticoagulants (e.g. warfarin, enoxaparin, or DOAC) within 14 days of study bronchoscopy
* Any symptoms consistent with infection including fever, chills, night sweats, or unexplained weight loss
* A history of a necrotic reaction to a tuberculin skin test, including during screening
* A history of human immunodeficiency virus (HIV) infection
* A history of coughing up blood in the last 3 months
* Cigarette smoking, vaping or recreational drug use within the past 6 months (self-reported)
* If there is any discrepancy in tuberculin skin test and Interferon Gamma Release Assay test results (i.e. PPD+ but IGRA- or PPD- but IGRA+)
* Refusal or inability to undergo bronchoscopy, or a history of poor tolerance of a bronchoscopy
* If undergoing PET-CT imaging during this study places a participant over his/her annual radiation dose limit. Radiation exposure within the previous 12 months of >= 2.3 rem
* BMI > 40
* Diabetes
* Known life-threatening allergic reaction to Tuberculin, Lidocaine, Midazolam, Fentanyl or medications of similar classes
* Presence of any immunosuppressive diseases, including cancers with the exception of non-melanomatous skin cancer.
* Use of any systemic immunosuppressive medications, including corticosteroids (e.g., prednisone) or biological agents in the last 6 months prior to enrollment
* Any medical, psychiatric, social condition, occupational reason or other responsibility, in the judgement of the investigator, that is a contraindication to protocol participation or impairs a participant s ability to give informed consent
* Positive for COVID-19. (with-in 6 months prior to enrollment self-reported and or via PCR)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Fennelly, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant results data will be made available 6 months after publication date for a period of 5 year by sending a request to kevin.fennelly@nih.gov
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available 6 months after publication date for a period of 5 year
Access Criteria: Sending request to kevin.fennelly@nih.gov

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-H-0027.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Healthy Volunteer Participants With Confirmed Latent Tuberculosis Infection (LTBI) | Arm 2: Healthy Volunteer Participants With Confirmed Non-Latent Tuberculosis Infection (LTBI)
Started | 7 | 10
Completed | 4 | 4
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non-compliance (missed one or more study visits) | 1 | 0
Not completed — Physician Decision | 1 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Healthy Volunteer Participants With Confirmed Latent Tuberculosis Infection (LTBI) | Arm 2: Healthy Volunteer Participants With Confirmed Non-Latent Tuberculosis Infection (LTBI) | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Median Difference in CD4 Cell Response to Intrabronchial Instillation of Tuberculin Purified Protein Derivative (PPD)
Description: Median difference in CD4 cell response to intrabronchial instillation of Tuberculin Purified Protein Derivative (PPD) using flow cytometry. The frequency of (Mycobacterium tuberculosis) Mtb-specific T cells was measured by intracellular cytokine staining for Interferon Gamma (IFNγ) and Tumor Necrosis Factor (TNF) after in vitro restimulation of Peripheral Blood Mononuclear Cells (PBMC) and Bronchoalveolar Lavage (BAL) cells with PPD or Mtb-derived peptide megapools.
Time Frame: Day 5 and Day 21
Population: Cryo-recovery of cells obtained from one participant was unsuccessful; therefore, analysis could not be performed.
Measure: Median (Inter-Quartile Range); unit: % Antigen Specific T cells
Arm/Group | Arm 1: Healthy Volunteer Participants With Confirmed Latent Tuberculosis Infection (LTBI) | Arm 2: Healthy Volunteer Participants With Confirmed Non-Latent Tuberculosis Infection (LTBI)
Number analyzed (Participants) | 4 | 4
% Antigen Specific T cells
  Day 5 | 5.26 [3.99 to 11.5] | 0.725 [0.462 to 1.74]
  Day 21: number analyzed (Participants) | 3 | 4
  Day 21 | 29.9 [19 to 37.3] | 2.92 [1.98 to 4.16]
Statistical Analysis 1: Comparison: Arm 1: Healthy Volunteer Participants With Confirmed Latent Tuberculosis Infection (LTBI) vs Arm 2: Healthy Volunteer Participants With Confirmed Non-Latent Tuberculosis Infection (LTBI); Test type: Superiority; p = 0.05714, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Median Difference in the Standard Uptake Value (SUV)
Description: Median difference in the Standard Uptake Value (SUV) in the pulmonary parenchyma and thoracic lymph nodes with positron emission tomography combined with chest computed tomography (PET-CT)
Time Frame: Baseline (Up to -7 days prior to PPD instillation), Day 4 and Day 20
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 30 Days
Description: At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization via in person, telephone and or e-mail.
Arm/Group | Arm 1: Healthy Volunteer Participants With Confirmed Latent Tuberculosis Infection (LTBI) | Arm 2: Healthy Volunteer Participants With Confirmed Non-Latent Tuberculosis Infection (LTBI)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 5/7 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Healthy Volunteer Participants With Confirmed Latent Tuberculosis Infection (LTBI) (N=7) | Arm 2: Healthy Volunteer Participants With Confirmed Non-Latent Tuberculosis Infection (LTBI) (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (2)
Red eyes (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bruising (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 1 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Injection site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Basophil count increased (Investigations) | 1 (1) | 0 (0)
C-Reactive Protein increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 3 (4)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Gag reflex (Nervous system disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Adnexal cystic mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (11) | 5 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidations (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paratracheal and suprahilar nodes (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (14) | 3 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema, upper arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Erythema, upper back (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (16) | 3 (16)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05027958/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT05027958/ICF_000.pdf